CLINICAL TRIAL: NCT06382025
Title: The Effect of Storybook vs Standart Information on Anesthesia Anxiety in Preoperative Period in Pediatric Patients
Brief Title: Preoperative Information With Storybook for Pediatric Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Trakya University (Other)
Responsible Party: Principal Investigator, Alkin Colak, Associate Professor, Trakya University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Alkinstorybook
Record Dates: First submitted 2024-04-15; First posted 2024-04-24 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Animation, Cartoons, Preoperative Care, Anesthesia, Pediatric

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- storybook (Active Comparator)
  Interventions: Other: showing cartoons -storybook
- standart (Placebo Comparator)
  Interventions: Other: showing cartoons - standard

INTERVENTIONS:
Other: showing cartoons -storybook — A goal-oriented 8-9 minutes animation cartoon that is informative and educational had been developed, and pediatric surgery patients had been asked to watch this animation during preoperative period
  Arms: storybook
Other: showing cartoons - standard — standard
  Arms: standart

SUMMARY:
Impacts of non-pharmacologic methods that help patients get prepared cognitively for processes of surgery and anesthesia on pediatric surgery patients' preoperational stress levels and anxiety levels had been examined in the scope of this comprehensive research project. In this project, a goal-oriented 8-9 minutes animation cartoon that is informative and educational had been developed, and pediatric surgery patients had been asked to watch this animation during preoperative period.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric surgery patient including inguinal hernia repair, circumcision and tonsillectomy.
* without having previous emergency surgery and anesthetic experience,

Exclusion Criteria:

* Their parents reported developmental delays, mental retardation, or chronic illnesses of the children
* Emergency surgery

Ages: 5 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 168 (Actual)
Dates: Start 2018-03-09 (Actual); Primary Completion 2020-02-20 (Actual); Study Completion 2020-05-29 (Actual)

PRIMARY OUTCOMES:
preoperative anxiety scale | baseline ( before induction of anesthesia)
State-trait anxiety inventory (STAI FORM TX-1, TX-2) for parents | baseline ( before induction of anesthesia)
Children's Hospital of Eastern Ontario Pain (CHEOP) Scale | Postoperative 0-24 hours
Pediatric Anesthesia Emergence Delirium (PAED) scale | Postoperative 1 hour

CONTACTS AND LOCATIONS:
Locations (1):
- Trakya University, Edirne, Edi̇rne, Turkey (Türkiye)